CLINICAL TRIAL: NCT03740282
Title: Prospective Clinical StuDy of Tri-planar Tarsometatarsal (TMT) ArthroDesIs With Early WeiGht-BeariNg After Lapiplasty ProcDure (ALIGN3D)
Brief Title: Early Weight-Bearing After the Lapiplasty Procedure
Acronym: ALIGN3D
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Treace Medical Concepts, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP2018-1
Record Dates: First submitted 2018-11-07; First posted 2018-11-14 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Hallux Valgus; Bunion
Keywords: arthrodesis; bunion; early weight-bearing; lapidus; hallux valgus
MeSH Terms: conditions — Hallux Valgus; Bunion; Ankylosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Lapiplasty (Experimental): All study participants receiving Lapiplasty procedure
  Interventions: Device: Lapiplasty

INTERVENTIONS:
Device: Lapiplasty — Patients 14 years through 58 years with symptomatic hallux valgus who are treated with the Lapiplasty System will begin weight-bearing by 3 weeks and follow a defined post-operative protocol.

SUMMARY:
The objectives of this study are to evaluate the following outcomes of the Lapiplasty® Procedure for patients in need of hallux valgus surgery:

* The study will determine the radiographic recurrence of hallux valgus and the timing of failure following hallux valgus correction with the Lapiplasty® Procedure.
* The study will determine whether the Lapiplasty® Procedure effectively corrects anatomical alignment of the 1st metatarsal and sesamoids in all three planes.
* The study will assess whether early weight-bearing after the Lapiplasty® Procedure affects the union rates or causes loss of 3-plane correction.
* The study will evaluate the quality of life and pain scores following the Lapiplasty® Procedure.

DETAILED DESCRIPTION:
Each subject will undergo the Lapiplasty® Procedure. The key surgical steps of the Lapiplasty® Procedure are releasing the 1st TMT joint, anatomical correction of the 3-plane deformity, bone preparation using the Lapiplasty® Cut Guide , provisional fixation and multiplanar permanent fixation with the BIPLANAR™ Plate.

It is common for people who undergo a Lapidus Arthrodesis to be non-weight-bearing for 6-8 weeks following the surgical procedure. This time allows the bones to properly fuse together. During this 6-8 week period, people can be limited in the typical day-to-day activities they participate in, such as walking, shopping and working.

The Lapiplasty® System Implants may allow subjects to bear weight earlier than traditional procedures without negatively effecting healing/union of the joint. By allowing people to bear weight earlier than traditional methods, it is possible that people will have the opportunity to resume typical day-to-day activities faster than usual.

This study will investigate the Lapiplasty® Procedure and the Lapiplasty® System Implants with early weight-bearing. The study preference is that subject will be placed in a walking CAM boot and allowed to start protected weight bearing no later than 3 weeks after surgery. Subject can begin protected bearing weight in a CAM boot as early as the day of surgery. Subject will return to weight-bearing in shoe (running or another athletic shoe) and full unrestricted activity as directed by the physician based on the clinical stability and subject ability to safely begin weight-bearing and unrestricted activities.

Recommended Approach for Post-Operative Care and Weight-Bearing Instructions

* Subject may be either bandaged, put in splint/cast or put in CAM boot at the time of surgery. If subject is fitted with CAM boot at discharge, the patient should be provided instructions on how to begin protected weight-bearing.
* Subject is instructed to remain off the operative foot as much as possible for the first few days post-op. This is to limit bleeding and swelling and to allow soft tissues to recover.
* Subject may leave the surgery facility with crutches, walker, rolling knee scooter or wheelchair.
* At the first post-op visit (0-3 weeks), bandages are removed, and the subject can be allowed to shower. Subject may wear an athletic sock. No bandages or splints are needed. The subject should be reminded of post-op care of the foot/surgical site.
* At the first post-op visit (0-3 weeks), the subject is fitted with a CAM boot (if the subject was not fitted for a CAM boot at discharge). Subject should be provided with instructions on how to begin protected weight-bearing in the CAM boot and acceptable activities:

  * Patient is instructed to put weight on foot as tolerated in the restrictive boot.
  * Patient is instructed not to roll forward onto the big toe and should remain on flat foot.
  * Patient is instructed to remove the CAM boot multiple times daily and perform range of motion exercises for ankle and foot.
* At the 6 week post-op visit, if the subject is clinically stable, subject can transition from the boot to a shoe (running or another athletic shoe). The transition from boot to shoe may occur over a period of days/weeks, depending on subject healing and tolerance. Subject is instructed that they can walk normally but are not to stand on toes, run, jump or do any other high impact activity
* At the 4 month post-op visit, subject is allowed to begin low impact exercise if they are clinically stable.

ELIGIBILITY:
Inclusion Criteria:

* Male and females between the ages 14 and 58 years at the time of consent
* Closed physeal plates at the time of consent
* Intermetatarsal angle is between 10.0 ̊ - 22.0 ̊
* Hallux valgus angle is between 16.0 ̊ - 40.0 ̊
* Willing and able to adhere to early weight-bearing instructions post-operatively
* Capable of completing self - administered questionnaires
* Acceptable surgical candidate, including use of general anesthesia
* Female patients must be of non-child bearing potential or have a negative pregnancy test within 7 days prior to index procedure
* Willing and able to schedule index procedure within 3 months of consent and able to return for scheduled follow-up visits
* Willing and able to provide written informed consent

Exclusion Criteria:

* Previous surgery for hallux valgus on operative side
* Previous surgeries on operative foot involving fusion of foot or ankle joints (other than hammertoe or lesser toes/digits)
* Additional arthrodesis outside the first tarsometatarsal joint (other than: arthrodesis between the medial cuneiform and intermediate cuneiform and/or base of 2nd metatarsal; arthrodesis of hammertoe proximal interphalangeal joint or lesser toes/digits)
* Moderate or Severe osteoarthritis of the MTP joint based on radiographic imaging (including lack of evident crista) or positive grind test
* Symptomatic flatfoot or asymptomatic flatfoot (defined as calcaneal inclination <5 ̊and talonavicular subluxation/uncovering >50%)
* BMI >40 kg/m²
* Current nicotine user, including current use of nicotine patch
* Current clinical diagnosis of diabetes with fasting plasma glucose > 126 mg/dL and/or HbA 1c ≥7.0
* Current clinical diagnosis of peripheral neuropathy or by assessment on 4 - point monofilament test
* Current clinical diagnosis of fibromyalgia
* Current clinical diagnosis of Complex Regional Pain Syndrome/Reflex Sympathetic Dystrophy (CRPS/RSD)
* Current uncontrolled hypothyroidism
* Previously sensitized to titanium
* Currently taking oral steroids or rheumatoid biologics
* Currently taking immunosuppressant drugs
* Insufficient quantity or quality of bone to permit stabilization, conditions that retard healing (not including pathological fractures) and conditions causing poor blood supply such as peripheral vascular disease
* Active, suspected or latent infection in the affected area
* Use of synthetic or allogenic bone graft substitutes
* Current diagnosis of metatarsus adductus (defined as MAA ≥ 23 ̊)
* Scheduled to undergo a same - bilateral procedure. Patient agrees to refrain from the Lapiplasty® Procedure (or other hallux valgus procedures) on contralateral foot for minimum of 6 months post index procedure
* Patient has previously been enrolled into this study for a contralateral procedure
* Scheduled for any concomitant procedure that would alter patient's ability to early weight-bear post-procedure
* Patient is actively involved with a workman's compensation case or is currently involved in litigation
* Patient is currently or has participated in a clinical study in the last 30 days prior to signing
* Patient has a condition or finding that, in the opinion of the Investigator, may jeopardize the patient's well-being, the soundness of this clinical study, or could interfere with provision of informed consent, completion of tests, therapy, or follow-up

Ages: 14 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 183 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Radiographic recurrence of hallux valgus | 24 Months
  Defined as IMA ≥ 12, HVA ≥ 20 and TSP as ≥ 4 at 24 Months post Lapiplasty Procedure

SECONDARY OUTCOMES:
Change in radiographic angular/positional alignment before and after the Lapiplasty Procedure | Pre-operatively, 6 Weeks, 4 Months, 6 Months, 12 Months, 24 Months, 36 Month, 48 Months, 60 Months
  Intermetatarsal Angle (IMA), Hallux Valgus Angle (HVA) and Tibial Sesamoid Position (TSP)
Clinical/radiographic healing | 12 Months
  Evaluate clinical/radiographic healing (union vs non-union). Non-union defined as lucency at TMT joint, hardware failure and/or loss of correction, plus clinical pain at first TMT joint at 12 Months post-Lapiplasty Procedure
Clinical complications | 24 Months
  Complications due to the Lapiplasty procedure device or post-operative protocol or health conditions that could affect other health outcomes
Time to start of weight-bearing in boot | 0-3 Weeks
  The time needed for a study subject to begin bearing weight in a boot after the Lapiplasty Procedure
Time to start of weight-bearing in shoes | 0-12 Weeks
  The time needed for a study subject to begin bearing weight in a shoe after the Lapiplasty Procedure
Time to return to full unrestricted activity | 6 Weeks to 12 Months
  The time needed for a study subject to return to full unrestricted activity after the Lapiplasty Procedure
Change in Visual Analog Scale (VAS) Pain Score | Pre-operatively, 6 Weeks, 4 Months, 6 Months, 12 Months, 24 Months, 36 Month, 48 Months, 60 Months
  Patient reported foot pain intensity/0 (no pain) - 10 (worst possible pain)
Change in PROMIS-29 score across multiple time-points | Pre-operatively, 6 Months, 12 Months, 24 Months
  Patient-Reported Outcomes Measurement Information System (PROMIS-29 Profile v2.1)/lowest possible score 29 - highest possible score 145. High scores mean more of the concept being measured.
Change in PROMIS-25 score across multiple time-points | Pre-operatively, 6 Months, 12 Months, 24 Months
  Patient-Reported Outcomes Measurement Information System (PROMIS-25 Profile v2.0)/lowest possible score 25 - highest possible score 135. High scores mean more of the concept being measured.
Change in MOxFQ Foot Problems score across multiple time-points | Pre-operatively, 6 Months, 12 Months, 24 Months
  Manchester-Oxford Foot Questionnaire (MOxFQ)/0 (minimum raw score) - 64 (maximum raw score). Raw score is converted to a metric of 0 - 100 with higher score representing greater severity
Change in Range of Motion | 12 Months, 24 Months
  1st MTP dorsiflexion and 1st MTP plantarflexion

CONTACTS AND LOCATIONS:
Overall Officials: Dane Wukich, MD, Principal Investigator — UTSW
Locations (7):
- United States (7):
  - Foot & Ankle Center of Northern Colorado, Greeley, Colorado
  - Foot & Ankle Center of Iowa, Ankeny, Iowa
  - Jefferson City Medical Group, P.C., Jefferson City, Missouri
  - Desert Orthopaedic Center, Las Vegas, Nevada
  - University of Pennsylvania/Penn Medicine, Philadelphia, Pennsylvania
  - UT Southwestern, Dallas, Texas
  - Stonebriar Foot & Ankle, Frisco, Texas

IPD SHARING:
Plan to Share IPD: No